CLINICAL TRIAL: NCT07210736
Title: Evolution of Neonates With Esophageal Atresia in Brazil - A Multicenter Study
Brief Title: Brazilian Multicenter Study on Esophageal Atresia
Acronym: NEOBRA-EA
Status: Not yet recruiting | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Ana Cristina Aoun Tannuri, Full professor, University of Sao Paulo General Hospital
Other Study IDs: 85624924.8.1001.0068
Record Dates: First submitted 2025-09-19; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Atresia
Keywords: Esophageal atresia; Surgical outcomes; Multicenter; Brazil
MeSH Terms: conditions — Esophageal Atresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group: Neonates diagnosed with esophageal atresia (with or without tracheoesophageal fistula) admitted to one of 72 participating neonatal centers in Brazil between January 2025 and December 2026. Eligible patients include those born in, or transferred to, a participating center within the first 15 days of life. All patients will be managed according to the treating institution's standard clinical and surgical practice.

SUMMARY:
Esophageal atresia is a congenital malformation where the esophagus does not form properly, often associated with a tracheoesophageal fistula. This condition requires complex surgical treatment and intensive neonatal care. Survival has improved worldwide, but results from other countries cannot be directly applied to Brazil due to differences in health resources. This study will gather data from 72 neonatal centers across Brazil to better understand the characteristics, treatments, complications, and outcomes of newborns with esophageal atresia. The goal is to identify factors associated with complications and mortality, and to generate national evidence that can guide better care and improve survival and quality of life.

DETAILED DESCRIPTION:
Esophageal atresia is a congenital malformation characterized by an interruption of the esophageal lumen, frequently associated with a tracheoesophageal fistula. Although survival has significantly improved over the past decades in high-income countries, outcomes remain heterogeneous, and the results from international registries cannot be directly extrapolated to the Brazilian context due to regional differences in health system resources, neonatal intensive care, and surgical practice. At present, Brazil lacks a comprehensive national study evaluating the epidemiology, management, and outcomes of neonates with esophageal atresia.

The present multicenter project represents the first nationwide collaboration dedicated to this condition. Seventy-two neonatal centers across Brazil will contribute data, creating a large national cohort that encompasses both retrospective and prospective cases.

Data collection will be standardized and managed using the REDCap platform (Research Electronic Data Capture), with local entry validated centrally at the coordinating center. Variables collected will include prenatal and perinatal information, associated anomalies, anatomical classification of the atresia, diagnostic procedures performed, intraoperative surgical details, postoperative course, complications, and mortality. Particular attention will be given to factors such as prematurity, congenital heart disease, VACTERL association, and "long-gap" esophageal atresia, as these conditions are expected to have significant impact on outcomes.

The study aims to describe the current Brazilian panorama of esophageal atresia, focusing on short- and mid-term outcomes, including mortality within the first year of life, early complications such as anastomotic leakage and sepsis, and late complications including strictures and recurrent fistulas. A multivariate statistical analysis will be performed to identify predictors of adverse outcomes and to compare the results of different treatment strategies adopted across participating centers.

This initiative is expected to provide unprecedented epidemiological and clinical insights into esophageal atresia in Brazil. By combining the expertise and data of multiple neonatal units across diverse regions, the study will generate robust evidence to guide best practices, inform clinical guidelines, and support improvements in neonatal surgical care. Ultimately, the findings have the potential to improve survival and quality of life for Brazilian neonates affected by this challenging congenital condition.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with a confirmed diagnosis of esophageal atresia of any anatomical type (with or without tracheoesophageal fistula).
* Birth in, or transfer to, one of the participating neonatal centers within the first 15 days of life.

Exclusion Criteria:

- Patients lost to follow-up before reaching 12 months of age.

Ages: 1 Minute to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will consist of neonates diagnosed with esophageal atresia admitted to 72 participating neonatal centers across Brazil. Eligible infants include those identified antenatally or perinatally and confirmed by clinical and diagnostic evaluation shortly after birth. Both term and preterm neonates will be included, and data on associated congenital anomalies will be collected.
  The cohort is designed to reflect the full clinical spectrum of esophageal atresia encountered in Brazilian neonatal surgical practice, including cases with distal fistula, isolated atresia without fistula, long-gap esophageal atresia, and patients with complex associated malformations such as congenital heart disease and VACTERL association.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality within the first year of life | From birth until 12 months of age
  Mortality from any cause in neonates with esophageal atresia, with or without tracheoesophageal fistula, who undergo standard surgical and neonatal management at participating centers. Mortality will include early deaths during initial hospitalization as well as late deaths up to 12 months of age.

SECONDARY OUTCOMES:
Surgical complications after primary repair of distal fistula | From surgery until 12 months of age
  Incidence of anastomotic dehiscence, stricture, and recurrent fistula among neonates with distal tracheoesophageal fistula undergoing primary surgical repair.
Incidence of postoperative complications among premature vs. term neonates with esophageal atresia | From birth until 12 months of age
  Number and percentage of neonates experiencing major postoperative complications (including anastomotic leakage, sepsis, stricture, or recurrent fistula) will be compared between premature (<37 weeks gestational age) and term infants.
Mortality rate among premature vs. term neonates with esophageal atresia | From birth until 12 months of age
  All-cause mortality will be compared between premature (<37 weeks gestational age) and term infants.
Incidence of postoperative sepsis among neonates with esophageal atresia | From surgery until 12 months of age
  Number and percentage of neonates experiencing postoperative sepsis will be reported. Sepsis will be defined according to Phoenix sepsis criteria for sepsis and septic shock.
Incidence of postoperative complications among neonates with long-gap esophageal atresia | From surgery until 12 months of age
  Number and percentage of neonates with long-gap esophageal atresia experiencing major postoperative complications (including anastomotic leakage, sepsis, stricture, or recurrent fistula) will be reported.
Incidence of mortality among neonates with long-gap esophageal atresia | From surgery until 12 months of age
  Number and percentage of neonates with long-gap esophageal atresia who die within 12 months after surgery will be reported.
Incidence of complications among neonates with vs. without associated congenital anomalies (cardiac or VACTERL components) | From birth until 12 months of age
  Number and percentage of neonates experiencing major postoperative complications will be compared between those with congenital anomalies (cardiac malformations or VACTERL association) and those without.
Mortality rate among neonates with vs. without associated congenital anomalies (cardiac or VACTERL components) | From birth until 12 months of age
  All-cause mortality will be compared between neonates with congenital anomalies (cardiac malformations or VACTERL association) and those without.

CONTACTS AND LOCATIONS:
Overall Officials: Ana C Tannuri, MD, PhD, Principal Investigator — Hospital das Clínicas HCFMUSP
Locations (1):
- Instituto da Crianca e do Adolescente, Hospital das Clinicas, Faculdade de Medicina, Universidade de Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ishimaru T, Fujiogi M, Michihata N, Matsui H, Fushimi K, Kawashima H, Fujishiro J, Yasunaga H. Impact of congenital heart disease on outcomes after primary repair of esophageal atresia: a retrospective observational study using a nationwide database in Japan. Pediatr Surg Int. 2019 Oct;35(10):1077-1083. doi: 10.1007/s00383-019-04542-w. Epub 2019 Aug 8. PMID 31396739
- [Background] Lal DR, Gadepalli SK, Downard CD, Ostlie DJ, Minneci PC, Swedler RM, Chelius TH, Cassidy L, Rapp CT, Billmire D, Bruch S, Burns RC, Deans KJ, Fallat ME, Fraser JD, Grabowski J, Hebel F, Helmrath MA, Hirschl RB, Kabre R, Kohler J, Landman MP, Leys CM, Mak GZ, Raque J, Rymeski B, Saito JM, St Peter SD, von Allmen D, Warner BW, Sato TT; Midwest Pediatric Surgery Consortium. Challenging surgical dogma in the management of proximal esophageal atresia with distal tracheoesophageal fistula: Outcomes from the Midwest Pediatric Surgery Consortium. J Pediatr Surg. 2018 Jul;53(7):1267-1272. doi: 10.1016/j.jpedsurg.2017.05.024. Epub 2017 Jun 1. PMID 28599967
- [Background] Tannuri U, Maksoud-Filho JG, Tannuri AC, Andrade W, Maksoud JG. Which is better for esophageal substitution in children, esophagocoloplasty or gastric transposition? A 27-year experience of a single center. J Pediatr Surg. 2007 Mar;42(3):500-4. doi: 10.1016/j.jpedsurg.2006.10.042. PMID 17336187
- [Background] Foker JE, Kendall TC, Catton K, Khan KM. A flexible approach to achieve a true primary repair for all infants with esophageal atresia. Semin Pediatr Surg. 2005 Feb;14(1):8-15. doi: 10.1053/j.sempedsurg.2004.10.021. PMID 15770584
- [Background] Tobia A, Luque CG, Leitmeyer K, Dorling M, Chadha NK. Endoscopic treatment in pediatric patients with recurrent and H-type tracheoesophageal fistulas - A systematic review and meta-analysis. Int J Pediatr Otorhinolaryngol. 2023 May;168:111541. doi: 10.1016/j.ijporl.2023.111541. Epub 2023 Mar 31. PMID 37043961
- [Background] Koivusalo A, Pakarinen MP, Rintala RJ. Anastomotic dilatation after repair of esophageal atresia with distal fistula. Comparison of results after routine versus selective dilatation. Dis Esophagus. 2009;22(2):190-4. doi: 10.1111/j.1442-2050.2008.00902.x. Epub 2008 Dec 22. PMID 19207547
- [Background] Aslanabadi S, Jamshidi M, Tubbs RS, Shoja MM. The role of prophylactic chest drainage in the operative management of esophageal atresia with tracheoesophageal fistula. Pediatr Surg Int. 2009 Apr;25(4):365-8. doi: 10.1007/s00383-009-2345-7. Epub 2009 Mar 17. PMID 19290533
- [Background] Davenport M, Rothenberg SS, Crabbe DC, Wulkan ML. The great debate: open or thoracoscopic repair for oesophageal atresia or diaphragmatic hernia. J Pediatr Surg. 2015 Feb;50(2):240-6. doi: 10.1016/j.jpedsurg.2014.11.008. Epub 2014 Nov 7. PMID 25638610
- [Background] Spitz L. Esophageal atresia. Lessons I have learned in a 40-year experience. J Pediatr Surg. 2006 Oct;41(10):1635-40. doi: 10.1016/j.jpedsurg.2006.07.004. PMID 17011260
- [Background] Goyal A, Jones MO, Couriel JM, Losty PD. Oesophageal atresia and tracheo-oesophageal fistula. Arch Dis Child Fetal Neonatal Ed. 2006 Sep;91(5):F381-4. doi: 10.1136/adc.2005.086157. PMID 16923940
- [Background] Roberts K, Karpelowsky J, Fitzgerald DA, Soundappan SS. Outcomes of oesophageal atresia and tracheo-oesophageal fistula repair. J Paediatr Child Health. 2016 Jul;52(7):694-8. doi: 10.1111/jpc.13211. Epub 2016 May 20. PMID 27206060